CLINICAL TRIAL: NCT06153121
Title: Construct and Predictive Validity of an Upper Extremity Physical Performance Test Battery in Healthy Athletes: a Cross-sectional and Prospective Study
Brief Title: Validity of an Upper Extremity Physical Performance Test Battery in Healthy Athletes
Acronym: VAL_PPT_H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ONZ-2023-0320
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult tennis players (Experimental): tennis players between the age of 18 and 40
  Interventions: Other: Physical performance test - Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST); Other: Physical performance test - Seated Seated Single Arm Shot Put Test (SSASPT); Other: Physical performance test - Upper Limb Rotation Test (ULRT); Other: Physical performance test - Shoulder endurance test (SET); Other: Analytical test - Hand Grip Strength; Other: Analytical test - Shoulder Range of Motion (ROM); Other: PROM - Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES); Other: PROM - Competitive State Anxiety Inventory-2 (CSAI-2); Other: PROM - General elf-efficacy scale (GSES).
- Adult swimmers (Experimental): swimmers between the age of 18 and 40
  Interventions: Other: Physical performance test - Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST); Other: Physical performance test - Seated Seated Single Arm Shot Put Test (SSASPT); Other: Physical performance test - Upper Limb Rotation Test (ULRT); Other: Physical performance test - Posterior shoulder endurance test (PSET); Other: Analytical test - Shoulder Strength; Other: Analytical test - Hand Grip Strength; Other: Analytical test - Shoulder Range of Motion (ROM); Other: PROM - Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES); Other: PROM - Competitive State Anxiety Inventory-2 (CSAI-2); Other: PROM - General elf-efficacy scale (GSES).
- Adolescent tennis players (Experimental): tennis players between the age of 12 and 18
  Interventions: Other: Physical performance test - modified Closed Kinetic Chain Upper Extremity Stability Test (m-CKCUEST); Other: Physical performance test - Seated Seated Single Arm Shot Put Test (SSASPT); Other: Physical performance test - Upper Limb Rotation Test (ULRT); Other: Physical performance test - Shoulder endurance test (SET); Other: Analytical test - Shoulder Strength; Other: Analytical test - Hand Grip Strength; Other: Analytical test - Shoulder Range of Motion (ROM); Other: PROM - Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES); Other: PROM - Competitive State Anxiety Inventory-2 (CSAI-2); Other: PROM - General elf-efficacy scale (GSES).
- Adolescent swimmers (Experimental): swimmers between the age of 12 and 18
  Interventions: Other: Physical performance test - modified Closed Kinetic Chain Upper Extremity Stability Test (m-CKCUEST); Other: Physical performance test - Seated Seated Single Arm Shot Put Test (SSASPT); Other: Physical performance test - Upper Limb Rotation Test (ULRT); Other: Physical performance test - Posterior shoulder endurance test (PSET); Other: Analytical test - Shoulder Strength; Other: Analytical test - Hand Grip Strength; Other: Analytical test - Shoulder Range of Motion (ROM); Other: PROM - Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES); Other: PROM - Competitive State Anxiety Inventory-2 (CSAI-2); Other: PROM - General elf-efficacy scale (GSES).

INTERVENTIONS:
Other: Physical performance test - Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) — The test is performed in a pushup position with the hands placed 91.4 cm apart on strips of athletic tape. The person reaches with alternating hands across the body to touch the piece of tape under the opposing hand. The number of cross-body touches performed in 15 seconds is recorded. In total, three 15-s test trials were performed, with 45 s rest between each trial.
  Arms: Adult swimmers; Adult tennis players
Other: Physical performance test - modified Closed Kinetic Chain Upper Extremity Stability Test (m-CKCUEST) — The test is performed in a pushup position with the hands one half-arm span apart on strips of athletic tape. The person reaches with alternating hands across the body to touch the piece of tape under the opposing hand. The number of cross-body touches performed in 15 seconds is recorded. In total, three 15-s test trials were performed, with 45 s rest between each trial.
  Arms: Adolescent swimmers; Adolescent tennis players
Other: Physical performance test - Seated Seated Single Arm Shot Put Test (SSASPT) — Set up requires that the subject is placed in a seated position with their back against the wall, and a 2kg medicine ball held in a shot put position. When ready, the subject will perform a shot put motion to project the medicine ball as far as possible. The average of three trials is recorded for each arm.
Other: Physical performance test - Upper Limb Rotation Test (ULRT) — Participants starts in a modified (on elbows) push-up position. Participants are positioned next to a wall in order to allow the shoulder, the elbow epicondyle, the greater trochanter and the lateral malleolus of the ankle to touch the wall. Participants are asked to perform a trunk rotation, coupled with an external rotation of the shoulder in a 90°-90° position (90° abduction, 90° external rotation) touching the tape placed vertically on the wall as quickly as possible for 15 s. Finally, three 15-s test trials were performed, with 45 s rest between each trial.
Other: Physical performance test - Shoulder endurance test (SET) — Participants were instructed to stand up straight with their back against a wall. The tested arm was placed in a 90°forward flexion holding a 1-m long thera-band® fixed at shoulder height on a graduated stick. Participants were asked to pull the thera-band® from the starting position 90°forward flexion-to a 90° external rotation and 90° abduction (90°90°position) at an alternated cadence given by a metronome. Males are asked to pull a green thera-band (2.1 kg) and females a red thera-band (1.7 kg). Repetitions are performed until the participant is fatigued.
  Arms: Adolescent tennis players; Adult tennis players
Other: Physical performance test - Posterior shoulder endurance test (PSET) — The participant is positioned prone, with the test shoulder off the table and the arm perpendicular to the floor. A bar on a stick is adjusted for each patient and fixed at the point that the participant's shoulder reaches 90° of horizontal abduction, the point at which the participant was to hold the arm at the top of the arc of motion for 1 second. The participant held a weight equal to 2% of his body weight (rounded to the nearest 0.5 kg). Starting with the arm perpendicular to the floor, the participant horizontally abducted his arm to 90 degrees at a cadence of 30 beats per minute. Repetitions are performed until the participant is fatigued.
  Arms: Adolescent swimmers; Adult swimmers
Other: Analytical test - Shoulder Strength — shoulder external rotation and internal rotation measured with a hand held dynanometer
  Arms: Adolescent swimmers; Adolescent tennis players; Adult swimmers
Other: Analytical test - Hand Grip Strength — Hand grip strength measured with a JAMAR Hand Dynamometer
Other: Analytical test - Shoulder Range of Motion (ROM) — Passive external rotation in supine position with arm in 90° abduction - passive internal rotation in supine position with arm in 90° abduction.
Other: PROM - Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES) — The KJOC-SES survey is composed of ten 10-point questions to evaluate specifically the performance of overhead athletes, with the highest performance score of 100.
Other: PROM - Competitive State Anxiety Inventory-2 (CSAI-2) — The Competitive State Anxiety Inventory scale contains 27 items. It a psychometric scale that asks the volunteer to rate, on a 4-point Likert scale, their coping skills for sports performance.
Other: PROM - General elf-efficacy scale (GSES). — The GSES measures (10 statements) how a person deals with stressors/difficult situations in life. The scale is about a person's self-confidence that his or her actions are responsible for successful outcomes or, in other words, that one has control over challenging demands imposed by the environment.

SUMMARY:
This project comprises two studies; a cross-sectional study and a prospective study.

1. The cross-sectional study aims to develop and validate a new sport-specific test battery (PROMs, analytical and physical performance tests) in healthy tennis players and swimmers.The construct validity of this upper extremity test battery will be examined through two different methods.

   1. Firstly, the performance on the test battery will be correlated to sport performance (sprint time at 100m freestyle in swimming and serve speed/accuracy in tennis)
   2. Secondly, the correlation between test battery performance and upper limb/trunk kinematics in a tennis serve (measured via inertial measurement units (IMUs)) will be examined.
2. In the prospective study, the predictive validity of the test battery will be evaluated. Healthy swimmers and tennis players will be tested at baseline using the same test battery as mentioned above. The athletes will be followed for one year and new injuries will be recorded via a weekly questionnaire. Performance on the test battery will be associated with the incidence of musculoskeletal injuries.

DETAILED DESCRIPTION:
Upper extremity physical performance tests (PPTs) of the upper limb are physically challenging tests and are supposed to be sport-specific and mimic the sport specific movements or load.

Currently, there is no strong evidence for the validity of many upper extremity physical performance tests, although these tests are widely used in the return-to-sport phase after upper limb injuries. There is a clear need for a validating test physical performance tests.

Validation of these PPTs is possible in several ways, e.g. correlation to an analytical construct such as strength. However, it is important that these tests are sport-specific. For this reason, the correlation between physical performance tests on the one hand and sports performance (in swimming and tennis) and upper limb kinematics during a tennis serve on the other hand will be evaluated in this study. However, a single PPT is unlikely to correlate strongly with sport performance or tennis serve kinematics, as previous studies have shown a weak to moderate association when a single PPT was correlated with sport performance or another construct. Therefore, a cluster of tests will be assessed; four PPTs per sport and three analytical tests measuring strength and mobility of shoulder and hand, since these are the cornerstone of testing protocols in sports rehabilitation.

In addition, patient-reported outcome measures (PROMs), questionnaires that measure physical and psychosocial factors, are becoming increasingly important in sports. Recent studies show that these factors influence sports performance and rehabilitation outcomes. Therefore, these questionnaires can be very useful in the return-to-sport phase and injury risk screening. The PROMs that will be used in this study are the following: Kerlan-Jobe Orthopedic Clinic Shoulder and Elbow Score (KJOC-SES), Competitive State Anxiety Inventory-2 (CSAI-2) and the general self-efficacy scale.

To conclude, the test battery consists of PPTs, analytical tests (strength and mobility) and PROMs.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Play tennis or swim competitively, at least 3 hours per week (training + competition)

Exclusion Criteria:

* History of shoulder dislocation in dominant and/or nondominant shoulder
* History of upper extremity surgery
* At the moment of participation, participants should not report a substantial injury (defined by the Oslo Sports Trauma Research Centre questionnaire on health problems) in the past two months. A substantial injury is defined as a moderate or severe reduction in training volume or reduction in sports performance or complete inability to participate in sport as substantial injuries and illnesses.
* Neurological symptoms in any extremity
* Suffering from a systemic disease (such as diabetes, lupus, arthrosis,.. )

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Sports performance | Baseline
  For tennis players: serve performance test (12 serves), consisting of serve velocity and accuracy
  * serve velocity: Peak SV was measured with a Stalker Professional sports radar Pro II+
  * serve accuracy: serve accuracy is evaluated based on a scoring system. Two points are awarded if the serve lands in the target area (target of 2x2 m down the "T"), only one point when serving into the serve box, and balls landing outside the serve box results in zero points. The score of every individual serve was summed up to a total score of a maximum of 24 points.
    * the average velocity and the total accuracy score is used for analysis
  For swimmers: time on 100m freestyle during competition event is used for analysis
New musculoskeletal injuries | During the 1 year follow-up after baseline measurements
  New musculoskeletal injuries registered by the OSTRC-H2 (The Oslo Sports Trauma Research Center Questionnaire on Health Problems)

SECONDARY OUTCOMES:
Range of motion, velocity and acceleration of the upper extremity during the tennis serve | Baselline
  Range of motion, velocity and acceleration of the upper extremity (wrist, elbow, shoulder, trunk) measured with inertial measurement units (IMUs) during the tennis serve

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, Principal Investigator — University Ghent
Locations (1):
- Department of rehabilitation sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided